CLINICAL TRIAL: NCT03037476
Title: Personalized Health Assessment Related to Medications (Project PHARM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jason Kilmer, Associate Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001782; 3U01DA040219-04S1 (NIH)
Record Dates: First submitted 2017-01-05; First posted 2017-01-31 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Feedback, Psychological; Clinical Trial; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based PFI (Experimental): Participants randomized to the web-based PFI in Study 2 receive a 5 component Personalized Feedback Tool. The first component is presented immediately after the baseline survey and a link to each of the remaining 4 components is sent to participants spaced 1 to 2 weeks apart. The PFI components cover: 1) Stimulants, 2) Marijuana, 3) PSM and unwanted effects, 4) Academics, and 5) Alcohol. Each component is comprised of personalized feedback presented in text and graphic format, and each component includes links to tips for making changes if and when the participant is contemplating or ready to commit to change. These tips include general relapse prevention strategies, as well as information about the importance of regular class attendance, study habits, and sleep habits for academic success. General educational tips/strategies for time management, as well as tips for initiating behavior change are also included. Each component takes approximately 5-10 minutes to review.
  Interventions: Behavioral: Web-based PFI
- Assessment Only (Other): The Assessment Only group receives assessment on substance use, health behaviors, and academic behaviors at baseline, 6-month follow-up, and 12-month follow-up in Study 2.
  Interventions: Behavioral: Assessment Only

INTERVENTIONS:
Behavioral: Web-based PFI — A web-based 5 component Personalized Feedback Tool covering content on: 1) Stimulants, 2) Marijuana, 3) PSM and unwanted effects, 4) Academics, and 5) Alcohol.
  Arms: Web-Based PFI
Behavioral: Assessment Only — The Assessment Only condition receives assessment on substance use, health behaviors, and academic behaviors at baseline, 6 month follow-up, and 12 month follow-up.
  Arms: Assessment Only

SUMMARY:
This research will adapt an evidence based intervention for alcohol and other drugs and evaluate its efficacy on Prescription Stimulant Medication (PSM) misuse in a web-based format for use with college students who have misused PSMs.

DETAILED DESCRIPTION:
This project proposes to evaluate the efficacy of Screening and Brief Interventions (SBIs) for reducing college students' PSM misuse through two different routes of screening and intervention across 9 colleges and universities spanning the United States. The research will consist of studies designed to 1) conduct focus groups to refine feedback materials (Study 1); 2) Conduct screening through the Registrar's student lists and implement a randomized controlled trial (RCT) of a web-based PSM intervention at all sites (Study 2); and 3) Evaluate the impact of the COVID-19 pandemic using the Study 2 sample on non-medical use of prescription stimulants, prescription opiates, alcohol use, marijuana use, and other substances during the COVID-19 pandemic, and understand motives, access, mental health impacts, and college student and young adult experiences during this unprecedented 12 months.

Study 1 consists of conducting up to 5 focus groups of 8-12 people to elicit feedback regarding the Personalized Feedback Tool and make refinements prior to carrying out Study 2.

In Study 2, students from 9 college campuses are screened for past year PSM misuse. Those meeting study criteria are invited to complete a web-based baseline survey and are randomized to either receive the web-based personalized feedback intervention (PFI) or to assessment only control. Participants complete follow-up assessments at 6 and 12 months post-baseline to evaluate intervention efficacy. The investigators hypothesize that participants who receive the PFI will reduce PSM misuse assessed at 6 and 12 month follow-ups. The investigators further expect reductions in perceived benefits of PSM and perceived descriptive norms for PSM, and increases in use of alternative behaviors to support academic success, and expect these changes will mediate impacts on PSM use at follow-ups. Secondary effects of the intervention on alcohol and marijuana use are also anticipated, and these reductions are expected to partially mediate PSM outcomes. Finally, PSM motives and demographics as potential moderators of intervention efficacy will also be explored.

Lastly, in February of 2021, we received approval to modify the aims for Study 3 to evaluate the impact of the COVID-19 pandemic using the Study 2 sample. In an already consented, recruited, and well-characterized sample of high-risk young adults reporting poly-substance use (Study 2 participants, n=843), Study 3 aimed to describe changes in non-medical use of prescription stimulants, prescription opiates, alcohol use, marijuana use, and other substances during the COVID-19 pandemic, and understand motives, access, mental health impacts, and college student and young adult experiences during this unprecedented 12 months. Specifically, we intend to evaluate changes pre- and post-pandemic in non-medical use of PSM, non-medical use of prescription opioid medications (POM), alcohol use, and marijuana use, as well as mood utilizing Study 2 baseline and follow-up data, controlling for intervention condition and time since last assessment. We also will evaluate student status and living arrangement as moderators. The investigators hypothesize: (1) Young adults will report less PSM and less POM during the pandemic compared to pre-pandemic assessments, in part due to reduced ease of access and a change in motives for use; (2) Given previous findings that academic motives were 8 of the 9 most frequently endorsed reasons for PSM, and given perceptions that a move to virtual learning has been less academically challenging, we hypothesize that academic motives for PSM will decrease significantly during the pandemic compared to pre-pandemic; (3) Those no longer in school will report less PSM and less POM during the pandemic compared to pre-pandemic. (4) Those living at home will have decreased alcohol and marijuana use compared to pre-pandemic. Among those reporting current student status at the time of the new survey, we will be able to evaluate changes in motives for use, access, and academic pressure from baseline to present.

ELIGIBILITY:
Study 1 Inclusion Criteria:

* Provides consent to participate
* Currently enrolled as a student at one of the participating campuses
* Between 18-25 year olds
* Misuse of prescription stimulants in the past year

Study 1 Exclusion Criteria:

* There are no exclusion criteria other than not meeting inclusion criteria.

Study 2 Inclusion Criteria:

* Provides consent to participate
* Currently enrolled as a student at one of the participating campuses and in their second semester/quarter or later
* Has an anticipated graduation date at least 12 months into the future
* Between 18-25 year olds
* Misuse of prescription stimulants in the past year

Study 2 Exclusion Criteria:

* There are no exclusion criteria other than not meeting inclusion criteria.

Study 3 Inclusion Criteria:

* Provides consent to participate
* Previous participation as a Study 2 participant.

Study 3 Exclusion Criteria:

* There are no exclusion criteria other than not meeting inclusion criteria.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 843 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Web-Based PFI | Assessment Only
Started | 414 | 429
Completed | 351 | 383
Not Completed | 63 | 46
Not completed — Lost to Follow-up | 63 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Web-Based PFI | Assessment Only | Total
Number analyzed (Participants) | 414 | 429 | 843
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45 | 31 | 76
  Between 18 and 65 years | 369 | 398 | 767
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.82 (1.12) | 19.95 (1.05) | 19.88 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 258 | 248 | 506
  Male | 156 | 181 | 337
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 41 | 87
  Not Hispanic or Latino | 366 | 388 | 754
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 81 | 88 | 169
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 21 | 16 | 37
  White | 263 | 276 | 539
  More than one race | 31 | 32 | 63
  Unknown or Not Reported | 15 | 11 | 26
Region of Enrollment [Number; unit: participants]
  United States | 414 | 429 | 843

OUTCOME MEASURES:

1. Primary Outcome: Change in Past 6 Month Non-Medical Use of Prescription Stimulant Medication Frequency
Description: Assesses frequency of non-medical use of prescription stimulant medications. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: Change in past 6 month number of days of nonmedical prescription stimulant use.
Measure: Mean (Standard Deviation); unit: Usage days
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 336 | 361
Usage days
  6 Month Follow-up | -2.04 (5.72) | -1.72 (6.88)
  12 Month Follow-up: number analyzed (Participants) | 316 | 348
  12 Month Follow-up | -1.03 (7.91) | -.38 (11.45)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Changes from Baseline to 6 Month Follow-up Outcomes reported in this section; Test type: Other — General Linear Model; p = 0.03, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.235, 95% CI 2-sided [-.446 to -.023]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Changes from Baseline to 12 Month Follow-up reported in this section; Test type: Other — General Linear Model; p = 0.164, Mixed Models Analysis; Negative Binomial Regression; Slope = -.149, 95% CI 2-sided [-.360 to .061]

2. Primary Outcome: Change in Past 6 Month Medical Misuse of Prescription Stimulant Medication
Description: Assesses past 6 month medical misuse of prescription stimulant medication. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: These analyses were limited to individuals who reported a diagnosis of ADHD (n=62).
Measure: Mean (Standard Deviation); unit: Usage days
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 27 | 35
Usage days
  6 Month Follow-up | -.30 (.72) | -.03 (.62)
  12 Month Follow-up | -.19 (.74) | -.07 (.66)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in Medical Misuse of Prescription Stimulant Medication Among those with ADHD Diagnosis from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .603, Mixed Models Analysis; Poisson Regression; Slope = -.24, 95% CI 2-sided [-1.120 to .650]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in Medical Misuse of Prescription Stimulant Medication Among those with ADHD Diagnosis from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .465, Mixed Models Analysis; Poisson Regression; Slope = -.336, 95% CI 2-sided [-1.238 to .566]

3. Primary Outcome: Change in Tobacco, Alcohol, Prescription Medications, and Substance Use/Misuse Brief Screen/Assessment Tool (TAPS Tool)
Description: Assesses problematic use of tobacco, alcohol, prescription, and illicit drugs over the past year and 3 months. Response options included: 0= Never, 1= Less than Monthly, 2= Monthly, 3= Weekly, 4= Daily or Almost Daily. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: Difference in number analyzed by condition are due to differences in follow-up participation rates and/or items skipped by participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 333 | 359
Score on a scale
  Change in Past 12 Month Tobacco Use at 6 Month Followup | -.03 (1.22) | .06 (.98)
  Change in Past 12 Month Tobacco Use at 12 Month Followup: number analyzed (Participants) | 314 | 349
  Change in Past 12 Month Tobacco Use at 12 Month Followup | 0.15 (1.35) | 0.15 (1.18)
  Change in Past 12 Month Alcohol Use at 6 Month Followup: number analyzed (Participants) | 333 | 357
  Change in Past 12 Month Alcohol Use at 6 Month Followup | -.12 (.90) | -.02 (.83)
  Change in Past 12 Month Alcohol Use at 12 Month Followup: number analyzed (Participants) | 314 | 349
  Change in Past 12 Month Alcohol Use at 12 Month Followup | -.09 (.89) | -.1 (.93)
  Change in Past 12 Month Other Drug Use at 6 Month Followup | -.16 (1.14) | -.18 (1.08)
  Change in Past 12 Month Other Drug Use at 12 Month Followup: number analyzed (Participants) | 314 | 349
  Change in Past 12 Month Other Drug Use at 12 Month Followup | -.17 (1.25) | -.22 (1.22)
  Change in Past 12 Month Nonmedical Prescription Drug Use at 6 Month Followup | -.26 (.87) | -.24 (.91)
  Change in Past 12 Month Nonmedical Prescription Drug Use at 12 Month Followup: number analyzed (Participants) | 314 | 349
  Change in Past 12 Month Nonmedical Prescription Drug Use at 12 Month Followup | -.3 (.97) | -.28 (.92)
  Change in Past 3 Month Tobacco Use at 6 Month Followup: number analyzed (Participants) | 332 | 359
  Change in Past 3 Month Tobacco Use at 6 Month Followup | -.04 (.59) | 0 (.53)
  Change in Past 3 Month Tobacco Use at 12 Month Followup: number analyzed (Participants) | 314 | 349
  Change in Past 3 Month Tobacco Use at 12 Month Followup | -.05 (.61) | .01 (.56)
  Change in Past 3 Month Alcohol Use at 6 Month Followup: number analyzed (Participants) | 314 | 333
  Change in Past 3 Month Alcohol Use at 6 Month Followup | -.05 (.78) | -.1 (.80)
  Change in Past 3 Month Alcohol Use at 12 Month Followup: number analyzed (Participants) | 291 | 315
  Change in Past 3 Month Alcohol Use at 12 Month Followup | -.90 (.81) | -.19 (.92)
  Change in Past 3 Month Marijuana Use at 6 Month Followup | -.12 (.76) | -.04 (.77)
  Change in Past 3 Month Marijuana Use at 12 Month Followup: number analyzed (Participants) | 314 | 349
  Change in Past 3 Month Marijuana Use at 12 Month Followup | -.06 (.80) | -.09 (.87)
  Change in Past 3 Month Stimulant Use at 6 Month Followup | -.02 (.58) | -.08 (.61)
  Change in Past 3 Month Stimulant Use at 12 Month Followup: number analyzed (Participants) | 313 | 349
  Change in Past 3 Month Stimulant Use at 12 Month Followup | -.09 (.66) | -.11 (.70)
  Change in Past 3 Month Heroin Use at 6 Month Followup | .01 (.26) | .01 (.15)
  Change in Past 3 Month Heroin Use at 12 Month Followup: number analyzed (Participants) | 313 | 349
  Change in Past 3 Month Heroin Use at 12 Month Followup | .01 (.28) | -.01 (.15)
  Change in Past 3 Month Nonmedical Prescription Drug Use at 6 Month Followup | -.01 (.26) | -.04 (.35)
  Change in Past 3 Month Nonmedical Prescription Drug Use at 12 Month Followup: number analyzed (Participants) | 314 | 349
  Change in Past 3 Month Nonmedical Prescription Drug Use at 12 Month Followup | .04 (.41) | -.03 (.36)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in Past 12 Month Tobacco Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .486, Mixed Models Analysis; Negative Binomial Regression; Slope = -.059, 95% CI 2-sided [-.227 to .108]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in Past 12 Month Tobacco Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .942, Mixed Models Analysis; Negative Binomial Regression; Slope = .006, 95% CI 2-sided [-.160 to .172]
Statistical Analysis 3: Comparison: Web-Based PFI vs Assessment Only; Change in Past 12 Month Alcohol Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .552, Mixed Models Analysis; Poisson Regression; Slope = -.042, 95% CI 2-sided [-.180 to .097]
Statistical Analysis 4: Comparison: Web-Based PFI vs Assessment Only; Change in Past 12 Month Alcohol Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .608, Mixed Models Analysis; Poisson Regression; Slope = .037, 95% CI 2-sided [-.104 to .177]
Statistical Analysis 5: Comparison: Web-Based PFI vs Assessment Only; Change in Past 12 Month Other Drug Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .840, Mixed Models Analysis; Poisson Regression; Slope = .015, 95% CI 2-sided [-.130 to .160]
Statistical Analysis 6: Comparison: Web-Based PFI vs Assessment Only; Change in Past 12 Month Other Drug Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .927, Mixed Models Analysis; Poisson Regression; Slope = .007, 95% CI 2-sided [-.142 to .155]
Statistical Analysis 7: Comparison: Web-Based PFI vs Assessment Only; Change in Past 12 Month Nonmedical Prescription Drug Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .932, Mixed Models Analysis; Poisson Regression; Slope = -.010, 95% CI 2-sided [-.244 to .223]
Statistical Analysis 8: Comparison: Web-Based PFI vs Assessment Only; Change in Past 12 Month Nonmedical Prescription Drug Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .648, Mixed Models Analysis; Poisson Regression; Slope = -.057, 95% CI 2-sided [-.300 to 0.187]
Statistical Analysis 9: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Tobacco Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .702, Mixed Models Analysis; Poisson Regression; Slope = -.059, 95% CI 2-sided [-.363 to .245]
Statistical Analysis 10: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Tobacco Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .524, Mixed Models Analysis; Poisson Regression; Slope = -.100, 95% CI 2-sided [-.408 to .208]
Statistical Analysis 11: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Alcohol Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .913, Mixed Models Analysis; Poisson Regression; Slope = .008, 95% CI 2-sided [-.137 to .153]
Statistical Analysis 12: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Alcohol Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .676, Mixed Models Analysis; Poisson Regresision; Slope = .032, 95% CI 2-sided [-.117 to .181]
Statistical Analysis 13: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Marijuana Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .712, Mixed Models Analysis; Poisson Regression; Slope = -.035, 95% CI 2-sided [-.223 to .152]
Statistical Analysis 14: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Marijuana Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .956, Mixed Models Analysis; Poisson Regression; Slope = .005, 95% CI 2-sided [-.186 to 0.197]
Statistical Analysis 15: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Stimulant Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .446, Mixed Models Analysis; Poisson Regression; Slope = .149, 95% CI 2-sided [-.234 to .531]
Statistical Analysis 16: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Stimulant Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .793, Mixed Models Analysis; Poisson Regression; Slope = .055, 95% CI 2-sided [-.353 to .462]
Statistical Analysis 17: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Heroin Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .999, Mixed Models Analysis; Negative Binomial Regression; Slope = -.001, 95% CI 2-sided [-2.005 to 2.003]
Statistical Analysis 18: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Heroin Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p = .397, Mixed Models Analysis; Negative Binomial Regression; Slope = .999, 95% CI 2-sided [-1.312 to 3.310]
Statistical Analysis 19: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Nonmedical Prescription Drug Use from Baseline to 6 Month Followup; Test type: Other — General Linear Model; p = .303, Mixed Models Analysis; Negative Binomial Regression; Slope = .465, 95% CI 2-sided [-.419 to 1.349]
Statistical Analysis 20: Comparison: Web-Based PFI vs Assessment Only; Change in Past 3 Month Nonmedical Prescription Drug Use from Baseline to 12 Month Followup; Test type: Other — General Linear Model; p < .05, Mixed Models Analysis; Negative Binomial Regression; Slope = .939, 95% CI 2-sided [.128 to 1.751]

4. Primary Outcome: Change in Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) - Stimulants Only
Description: Measures past 3 month non-medical use of prescription stimulants and associated negative consequences. Items were summed to create a scale summary score where higher values indicated more problematic use in the past 3 months (min=0, max=40). Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 330 | 356
Score on a scale
  Change in ASSIST score at 6 month follow up | -1.420 (4.59) | -1.08 (5.02)
  Change in ASSIST score at 12 month follow up: number analyzed (Participants) | 312 | 344
  Change in ASSIST score at 12 month follow up | -1.26 (5.35) | -1.19 (5.24)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in ASSIST Score over time: 6 month follow up; Test type: Other — General Linear Model; p = 0.151, Mixed Models Analysis; Negative binomial regression; Slope = -0.1816, 95% CI 2-sided [-0.4295 to 0.0663]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Changes in ASSIST scores at 12 month follow up; Test type: Other — General Linear Model; p = 0.642, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0601, 95% CI 2-sided [-0.3133 to 0.1931]

5. Primary Outcome: Change in Past 6 Month Prescription Stimulant Use Consequence Questionnaire
Description: Assesses negative consequences associated with prescription stimulant misuse over the previous 6 months. A score of "0" indicates that a given consequence did not occur and a score of "1" indicates that it did occur. Items were summed to create a scale summary score of overall number of unique consequences that occurred in the past 6 months (min=0, max=19). Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: 6 and 12 month follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 329 | 357
Score on a scale
  Change in consequence score at 6 months | -1.27 (3.8) | -1.07 (3.65)
  Change in consequence score at 12 months: number analyzed (Participants) | 308 | 342
  Change in consequence score at 12 months | -0.92 (4.15) | -1.11 (4.16)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in consequence score at 6 month follow up; Test type: Other — General Linear Model; p = 0.074, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.2177, 95% CI 2-sided [-0.4566 to 0.0213]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in consequence score at 12 month follow up; Test type: Other — General Linear Model; p = 0.351, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.1165, 95% CI 2-sided [-0.3612 to 0.1282]

6. Secondary Outcome: Change in Peak Quantity of Alcohol Consumed in Past Month
Description: Assesses quantity in standard drinks of peak drinking episode of alcohol consumption over the past month. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 322 | 357
standard drinks
  Change in peak alcohol standard drink total at 6 months | -0.94 (3.71) | -1.23 (4.14)
  Change in peak standard drink total at 12 months: number analyzed (Participants) | 310 | 345
  Change in peak standard drink total at 12 months | -1.26 (3.82) | -1.48 (4.53)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in peak alcohol quantity at 6 months (reported by number of standard drinks); Test type: Other — General Linear Model; p = 0.255, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.0440, 95% CI 2-sided [-0.032 to 0.1197]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in peak alcohol quantity (reported in standard drinks) at 12 month follow-up; Test type: Other — General Linear Model; p = 0.428, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.0315, 95% CI 2-sided [-0.0463 to 0.1092]

7. Secondary Outcome: Change in Past 6 Month Daily Drinking Questionnaire
Description: Assesses typical alcohol consumption over the course of a typical week. Responses for number of drinks consumed each day of a typical week were summed to create a summary score of total number of drinks consumed over a typical week. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of drinks
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 312 | 350
Number of drinks
  Change in DDQ score at 6 months | -2.09 (6.92) | -2.11 (7.22)
  Change in DDQ score at 12 months: number analyzed (Participants) | 303 | 337
  Change in DDQ score at 12 months | -2.81 (8.60) | -2.07 (8.59)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in DDQ score at 6 months; Test type: Other — General Linear Model; p = 0.966, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.0021, 95% CI 2-sided [-0.0936 to 0.0978]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in DDQ score at 12 month follow-up; Test type: Other — General Linear Model; p = 0.265, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0559, 95% CI 2-sided [-0.1542 to 0.0424]

8. Secondary Outcome: Change in Past 6 Month Rutgers Alcohol Problem Index
Description: Measures negative alcohol-related consequences experienced over the past 6 months. A score of "0" indicates that a given consequence did not occur and a score of "1" indicates that it did occur. Items were summed to create a scale summary score of overall number of unique consequences that occurred in the past 6 months (min=0, max=26). Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 321 | 356
Score on a scale
  Change in RAPI score at 6 month follow up | -1.66 (5.06) | -1.42 (4.44)
  Change in RAPI score at 12 month follow up: number analyzed (Participants) | 304 | 342
  Change in RAPI score at 12 month follow up | -1.47 (5.71) | -1.21 (4.94)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in RAPI count at 6 month follow-up; Test type: Other — General Linear Model; p = 0.868, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0128, 95% CI 2-sided [-0.1633 to 0.1378]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in RAPI count at 12 month follow-up; Test type: Other — General Linear Model; p = 0.573, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0445, 95% CI 2-sided [-0.1993 to 0.1102]

9. Secondary Outcome: Change in Past Year, 6 Month, and 30 Day Marijuana Use Frequency
Description: Items measure typical frequency of marijuana use and number of days used in the past year, 6 months, and 30 days. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Usage days
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 320 | 353
Usage days
  Change in past year marijuana use at 6 month follow up | 2.22 (72.74) | 3.60 (66.67)
  Change in past year marijuana use at 12 month follow up: number analyzed (Participants) | 306 | 342
  Change in past year marijuana use at 12 month follow up | 3.90 (84.00) | 0.35 (87.60)
  Change in past 6 month marijuana use at 6 month follow-up | 0.49 (36.58) | 1.69 (34.04)
  Change in past 6 month marijuana use at 12 month follow-up: number analyzed (Participants) | 306 | 342
  Change in past 6 month marijuana use at 12 month follow-up | 2.22 (41.52) | -0.57 (42.00)
  Change in past month marijuana use at 6 month follow-up: number analyzed (Participants) | 319 | 353
  Change in past month marijuana use at 6 month follow-up | -0.07 (7.22) | 0.00 (7.33)
  Change in past month marijuana use at 12 month follow-up: number analyzed (Participants) | 305 | 342
  Change in past month marijuana use at 12 month follow-up | -0.53 (8.56) | -0.39 (8.47)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in past 12 month marijuana use at 6 month follow-up; Test type: Other — General Linear Model; p = 0.266, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0899, 95% CI 2-sided [-0.2484 to 0.0685]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Past 12 month marijuana use at 12 month follow-up; Test type: Other — General Linear Model; p = 0.816, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0197, 95% CI 2-sided [-0.1859 to 0.1465]
Statistical Analysis 3: Comparison: Web-Based PFI vs Assessment Only; Change in past 6 month marijuana use at 6 month follow-up; Test type: Other — General Linear Model; p = 0.209, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.1031, 95% CI 2-sided [-0.2639 to 0.0577]
Statistical Analysis 4: Comparison: Web-Based PFI vs Assessment Only; Change in past 6 month marijuana use at 12 month follow-up; Test type: Other — General Linear Model; p = 0.944, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0060, 95% CI 2-sided [-0.1729 to 0.1608]
Statistical Analysis 5: Comparison: Web-Based PFI vs Assessment Only; Change in past month marijuana use at 6 month follow-up; Test type: Other — General Linear Model; p = 0.654, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0391, 95% CI 2-sided [-0.2102 to 0.1320]
Statistical Analysis 6: Comparison: Web-Based PFI vs Assessment Only; Change in past month marijuana use at 12 month follow-up; Test type: Other — General Linear Model; p = 0.481, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0646, 95% CI 2-sided [-0.2444 to 0.1152]

10. Secondary Outcome: Change in Past 6 Month Rutgers Marijuana Problem Index
Description: Measures negative marijuana-related consequences experienced over the past 6 months. A score of "0" indicates that a given consequence did not occur and a score of "1" indicates that it did occur. Items were summed to create a scale summary score of overall number of unique consequences that occurred in the past 6 months (min=0, max=26). Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 316 | 347
Score on a scale
  Change in RMPI count at 6 month follow up | -0.81 (6.13) | -0.66 (5.53)
  Change in RMPI count at 12 month follow up: number analyzed (Participants) | 304 | 339
  Change in RMPI count at 12 month follow up | -0.81 (6.00) | -1.01 (6.20)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in RMPI count at 6 month follow-up; Test type: Other — General Linear Model; p = 0.487, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0411, 95% CI 2-sided [-0.1569 to 0.0747]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in RMPI count at 12 month follow-up; Test type: Other — General Linear Model; p = 0.772, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.0177, 95% CI 2-sided [-0.1021 to 0.1375]

11. Other Pre Specified Outcome: Change in Past 6 Month Relapse Prevention/Protective Behaviors Scale
Description: Measures the use of relapse prevention strategies and protective behaviors related to stimulant medication misuse. A score of "0" indicates that a given strategy did not occur and a score of "1" indicates that it did occur. Items were summed to create a scale summary score of overall number of unique relapse prevention/protective behavior strategies that occurred in the past 6 months (min=0, max=28). Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 316 | 347
Score on a scale
  Change in PBS count at 6 month follow up | -0.32 (6.03) | -1.40 (6.62)
  Change in PBS count at 12 month follow up: number analyzed (Participants) | 302 | 337
  Change in PBS count at 12 month follow up | -0.77 (7.36) | -1.30 (6.80)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in PBS count at 6 month follow up; Test type: Other — General Linear Model; p = 0.075, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.1285, 95% CI 2-sided [-0.0131 to 0.2702]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in PBS count at 12 month follow up; Test type: Other — General Linear Model; p = 0.207, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.0936, 95% CI 2-sided [-0.0517 to 0.2388]

12. Other Pre Specified Outcome: Change in Past Year Prescription Stimulant Norms Rating Form
Description: Assesses the perceived percentage of students who have misused prescription stimulant medication in the past year. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 336 | 360
Percentage
  Change in perceived norm (in perceived past year days of use) at 6 month | -9.29 (19.37) | -4.11 (20.44)
  Change in perceived norm (in perceived past year days of use) at 12 month: number analyzed (Participants) | 319 | 348
  Change in perceived norm (in perceived past year days of use) at 12 month | -11.10 (20.99) | -6.36 (18.50)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in perceived norm (in perceived days of use in past year) at 6 month follow up; Test type: Other — General Linear Model; p < 0.001, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.1604, 95% CI 2-sided [-0.2525 to -0.0683]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in perceived norm (perceived number of days of use in past year) at 12 month follow up; Test type: Other — General Linear Model; p < .003, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.1441, 95% CI 2-sided [-0.2404 to -0.0478]

13. Other Pre Specified Outcome: Change in Current Semester/Quarter Motivated Strategies for Learning Questionnaire (MSLQ)
Description: A 19-item abbreviated version of the Motivated Strategies for Learning Questionnaire was used to measures the use of different types of learning strategies and academic motivations during the current semester/quarter. Response options ranged from 1=Not at all true of me to 7=Very true of me. Mean scale scores were computed and change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 312 | 351
Score on a scale
  Change in MSLQ score at 6 month follow up | -0.10 (1.07) | -0.08 (0.95)
  Change in MSLQ score at 12 month follow up: number analyzed (Participants) | 295 | 338
  Change in MSLQ score at 12 month follow up | -0.01 (1.06) | -0.1 (1.09)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in MSLQ score at 6 month follow-up; Test type: Other — General Linear Model; p = 0.743, Mixed Models Analysis; Poisson regression; Slope = -0.0157, 95% CI 2-sided [-0.1096 to 0.0782]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in MSLQ score at 12 month follow up; Test type: Other — General Linear Model; p = 0.784, Mixed Models Analysis; Poisson regression; Slope = 0.0133, 95% CI 2-sided [-0.0816 to 0.1081]

14. Other Pre Specified Outcome: Change in Cumulative and Last Semester/Quarter Grade Point Average (GPA)
Description: Participants report their cumulative and previous semester/quarter GPA. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: 6 and 12 month follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 335 | 366
Score on a scale
  Change in cumulative GPA at 6 month follow up | 0.01 (0.21) | -0.002 (0.20)
  Change in cumulative GPA at 12 month follow-up: number analyzed (Participants) | 322 | 354
  Change in cumulative GPA at 12 month follow-up | 0.02 (0.26) | 0.03 (0.24)
  Change in last term GPA at 6 month follow-up: number analyzed (Participants) | 335 | 364
  Change in last term GPA at 6 month follow-up | 0.05 (0.45) | 0.01 (0.45)
  Change in last term GPA at 12 month follow-up: number analyzed (Participants) | 321 | 352
  Change in last term GPA at 12 month follow-up | 0.05 (0.50) | 0.24 (0.48)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in cumulative grade point average at 6 month follow up; Test type: Other — General Linear Model; p = 0.914, Mixed Models Analysis; Poisson regression; Slope = -0.0061, 95% CI 2-sided [-0.1161 to 0.104]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in cumulative grade point average at 12 month follow up; Test type: Other — General Linear Model; p = 0.871, Mixed Models Analysis; General Linear Model; Slope = -0.0092, 95% CI 2-sided [-0.1202 to 0.1018]
Statistical Analysis 3: Comparison: Web-Based PFI vs Assessment Only; Change in last term GPA at 6 month follow-up; Test type: Other — General Linear Model; p = 0.957, Mixed Models Analysis; Poisson regression; Slope = 0.0030, 95% CI 2-sided [-0.1063 to 0.1124]
Statistical Analysis 4: Comparison: Web-Based PFI vs Assessment Only; Change in last term GPA at 12 month follow-up; Test type: Other — General Linear Model; p = 0.992, Mixed Models Analysis; Poisson regression; Slope = 0.0006, 95% CI 2-sided [-0.1098 to 0.1109]

15. Secondary Outcome: Change in Frequency of Past Month Alcohol Consumption
Description: Assesses frequency (days) of alcohol consumption over the past month (min=0, max=31). Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Usage days
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 322 | 357
Usage days
  Change in past month frequency alcohol at 6 months | -1.21 (4.94) | -1.61 (5.45)
  Change in past month alcohol frequency at 12 months | -1.04 (5.63) | -1.30 (6.36)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in past month alcohol frequency at 6 month follow-up; Test type: Other — General Linear Model; p = 0.447, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.039, 95% CI 2-sided [-.0615 to 0.1395]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in past month alcohol frequency at 12 month follow-up; Test type: Other — General Linear Model; p = 0.443, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.0398, 95% CI 2-sided [-0.0619 to 0.1414]

16. Secondary Outcome: Change in Typical Quantity in Standard Drinks Consumed on a Typical Occasion in the Past Month
Description: Assesses typical drinking quantity in standard drinks of alcohol consumed during a typical drinking occasion over the past month. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline and the value at 12 months minus the value at baseline).
Time Frame: Baseline and 6 months, Baseline and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Web-Based PFI | Assessment Only
Number analyzed (Participants) | 322 | 357
standard drinks
  Change in past month typical quantity at 6 months | -1.47 (3.82) | -1.40 (3.89)
  Change in past month typical quantity at 12 months | -1.90 (4.16) | -1.57 (4.42)
Statistical Analysis 1: Comparison: Web-Based PFI vs Assessment Only; Change in past month alcohol typical quantity at 6 months; Test type: Other — General Linear Model; p = 0.997, Mixed Models Analysis; Negative Binomial Regression; Slope = 0.0002, 95% CI 2-sided [-0.1066 to 0.1070]
Statistical Analysis 2: Comparison: Web-Based PFI vs Assessment Only; Change in past month typical alcohol quantity at 12 month follow-up; Test type: Other — General Linear Model; p = 0.808, Mixed Models Analysis; Negative Binomial Regression; Slope = -0.0136, 95% CI 2-sided [-0.1236 to 0.0963]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Web-Based PFI | Assessment Only
All-Cause Mortality (participants affected / at risk) | 0/414 | 0/429
Serious Adverse Events (participants affected / at risk) | 0/414 | 0/429
Other Adverse Events (participants affected / at risk) | 0/414 | 0/429

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03037476/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03037476/ICF_001.pdf